CLINICAL TRIAL: NCT05273515
Title: The Acceptability and Feasibility of 3D Reconstruction and Virtual Reality in Addressing Body Image in Bariatric Surgery
Brief Title: Virtual Reality and 3D Reconstruction in Body Image and Bariatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 312801; 22IC7677 (Other: Imperial College London)
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Body Image Disorder; Bariatric Surgery Candidate
Keywords: Virtual Reality; 3D Reconstruction; Bariatric Surgery
MeSH Terms: conditions — Obesity; Body Dysmorphic Disorders

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot (Experimental): 3D scanning of participants. Images used to created 3D reconstruction of 15% and 25% total body weight loss. These are shown to participants using virtual reality. Qualitative outcomes measured using group discussion and questionnaires.
  Interventions: Other: Virtual Reality and 3D Reconstruction

INTERVENTIONS:
Other: Virtual Reality and 3D Reconstruction — Using virtual reality and 3D reconstruction to produce personalise images of what participants may look like after 15% and 25% total weight loss.

SUMMARY:
With obesity on the rise, the number of metabolic procedures performed annually is also increasing. Bariatric surgery has a significant impact on metabolic disease but also results in significant weight loss. Approximately, 30-40% of excess weight is lost within the first year following surgery. One of the motivating factors for surgery for patients is body image dissatisfaction and the stigmatisation of living with obesity, which is linked to low esteem, anxiety and depression. However, studies have indicated that following bariatric surgery, patients continue to experience dissatisfaction with their new body and identity due to unmet expectations.

The investigators aim is to start addressing body image issues prior to surgery and provide realistic expectations to patients. This study will be focusing on the feasibility and acceptability of 3D image reconstruction and virtual reality as a method of helping bariatric patients manage their expectations and improve body image satisfaction after surgery. Thereby, leading to better quality of life, improved psychological outcomes and prevention of disordered eating, anxiety and depression.

The study will take place at St Mary's Hospital (London) and the West London NHS Trust Bariatric Clinic from March 2022 to September 2022 (7 months). The study aims to recruit 10 participants from the Tier 3 Bariatric Preoperative Group. Once the participant has provided written consent, a photograph of them will be taken using a handheld 3D scanner on a secure password protected device. The images will be processed to produce two reconstructed images, one with 15% less body weight and the second with 25% less body weight. The participants will be divided into groups of 5 and shown their reconstructed images using individual virtual reality headsets. The participants will only have access to their own images. This will be followed up with group peer discussion meetings and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* In the tier 3 preoperative bariatric group
* 18 to 75 years old
* Male and Female

Exclusion Criteria:

* Anyone who cannot provide informed consent.
* Anyone with significant mental health instability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire to assess acceptability and Feasibility of Virtual Reality and 3d Reconstruction in Body Image and Bariatric Surgery | 6 months
  The primary outcome measure for the study is whether virtual reality and 3D reconstruction is an acceptable and feasible method of providing psychological support to bariatric patients. This will be determined from the responses on the feedback questionnaires. Participants will undertake 3 questionnaires; 1st after 15% less body weight image shown, 2nd after 25% less body weight image shown and 3rd after final peer group meeting.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bello, PhD, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study with only 10 participants, individual participant data will not be made available to other researchers. The results will be checked by the sponsor - Imperial College London

REFERENCES:
- [Background] Ionut V, Bergman RN. Mechanisms responsible for excess weight loss after bariatric surgery. J Diabetes Sci Technol. 2011 Sep 1;5(5):1263-82. doi: 10.1177/193229681100500536. PMID 22027328
- [Background] Bianciardi E, Di Lorenzo G, Niolu C, Betro S, Zerbin F, Gentileschi P, Siracusano A. Body image dissatisfaction in individuals with obesity seeking bariatric surgery: exploring the burden of new mediating factors. Riv Psichiatr. 2019 Jan-Feb;54(1):8-17. doi: 10.1708/3104.30935. PMID 30760932
- [Background] Legenbauer T, Muller A, de Zwaan M, Herpertz S. Body Image and Body Avoidance Nine Years After Bariatric Surgery and Conventional Weight Loss Treatment. Front Psychiatry. 2020 Jan 14;10:945. doi: 10.3389/fpsyt.2019.00945. eCollection 2019. PMID 31992997
- [Background] Ivezaj V, Grilo CM. The complexity of body image following bariatric surgery: a systematic review of the literature. Obes Rev. 2018 Aug;19(8):1116-1140. doi: 10.1111/obr.12685. Epub 2018 Jun 13. PMID 29900655
- [Background] Cruz-Saez S, Pascual A, Salaberria K, Etxebarria I, Echeburua E. Risky eating behaviors and beliefs among adolescent girls. J Health Psychol. 2015 Feb;20(2):154-63. doi: 10.1177/1359105313500683. Epub 2013 Sep 20. PMID 24058109
- [Background] Conceicao E, Orcutt M, Mitchell J, Engel S, Lahaise K, Jorgensen M, Woodbury K, Hass N, Garcia L, Wonderlich S. Eating disorders after bariatric surgery: a case series. Int J Eat Disord. 2013 Apr;46(3):274-9. doi: 10.1002/eat.22074. Epub 2012 Nov 29. PMID 23192683
- [Background] Caltabiano ML. Translational aspects of body image research for obesity-related quality of life and weight loss maintenance post-bariatric surgery. Ann Transl Med. 2020 Mar;8(Suppl 1):S2. doi: 10.21037/atm.2019.09.63. PMID 32309406
- [Background] Ratcliffe D, Ali R, Ellison N, Khatun M, Poole J, Coffey C. Bariatric psychology in the UK National Health Service: input across the patient pathway. BMC Obes. 2014 Aug 30;1:20. doi: 10.1186/s40608-014-0020-6. eCollection 2014. PMID 26217507
- [Background] Phelan S, Peruvemba S, Levinson D, Stulberg N, Lacy A, Legato M, Werner JP. Feasibility of a virtual reality-based approach to improve behavioral weight management outcomes. Pilot Feasibility Stud. 2021 Jun 22;7(1):129. doi: 10.1186/s40814-021-00865-5. PMID 34158129
- [Background] Manzoni GM, Cesa GL, Bacchetta M, Castelnuovo G, Conti S, Gaggioli A, Mantovani F, Molinari E, Cardenas-Lopez G, Riva G. Virtual Reality-Enhanced Cognitive-Behavioral Therapy for Morbid Obesity: A Randomized Controlled Study with 1 Year Follow-Up. Cyberpsychol Behav Soc Netw. 2016 Feb;19(2):134-40. doi: 10.1089/cyber.2015.0208. Epub 2015 Oct 2. PMID 26430819
- See also: Bariatric Surgery Register — https://e-dendrite.com/Publishing/Reports/Bariatric/NBSR2020.pdf